CLINICAL TRIAL: NCT00721240
Title: Investigation to Identify Predictors of Response to a Treatment With Montelukast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marien Hospital Wesel (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr. Andrea von Berg, Marien Hospital Wesel, Forschungsinstitut zur Prävention von Allergien und Atemwegserkrankungen im Kindesalter an der Klinik für Kinder- und Jugendmedizin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trial No. 25.08.2005
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2008-07

CONDITIONS: Asthma
Keywords: responder; leucotriene antagonist
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single-arm (Experimental): This investigation is a single-center, two-phase, single-arm study. In order to detect a potential placebo effect, the treatment phase will be preceded by a single-blinded two-week placebo run-in phase, followed by a 12 week open-label treatment phase.
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: montelukast — 5mg montelukast once daily for 12 weeks
  Other Names: Singulair ; MK-476

SUMMARY:
The main aim of the study is to develop a method that allows responders to be distinguished from non-responders before long-term treatment is initiated. Subsidiary aims are to record changes in pulmonary functional parameters, NO concentrations and peak flow variability, the use of beta2 sympathomimetics and the asthma symptom score.

DETAILED DESCRIPTION:
Leukotriene antagonists (montelukast) are particularly effective as controllers before exposure to an allergen (Leff 1998). The same applies to the treatment of bronchoconstriction induced by physical exertion or cold air (Richter 2000). Montelukast binds to the cysteinyl leuko¬triene-1 receptor, where it prevents leukotriene from binding. Leukotrienes play a key role as mediators in inflammatory processes. By binding to the receptor they cause, among other things, edema, damage to the bronchial epithelium and bronchoconstriction. Accordingly, in addition to its anti-inflammatory activity montelukast brings about bronchial dilation. The safety and efficacy of the drug in children have been well documented (Knorr 1998). Hence montelukast is approved for the treatment of bronchial asthma in children (over six months of age). As with other antiasthmatic drugs, there are responders and nonresponders to leukotriene receptor antagonists. The proportion of nonresponders to montelukast among children is esti¬mated to be 30% to 40%. At present the only way to distinguish non-responders from responders is to run a treatment trial for several weeks. If the symptom score falls, if the use of beta2 sympathomimetics is reduced, if pulmonary function and/or the quality of life improves, it is assumed that the patient is a responder. This method is not only tedious but also unsafe, since a change is the aforementioned parameters could occur spontaneously, without this being reliably attributable to the influence of the drug. In the planned study approximately 30 children with asthma of GINA classes 2 and 3 will be regularly examined for pulmonary function, symptom score and nitrogen monoxide (NO). First, however, the acute pharmacologic effect of a single dose of montelukast will be deter¬mined over a period of four hours by measuring pulmonary function and levels of exhaled nitrogen monoxide (NO).

4.2.1. Questions addressed:

Is it possible to discriminate between responders and nonresponders at a very early stage on the basis of the acute pharmacologic effect of montelukast? Does this classification agree with the results after 12 weeks of treatment?

4.2.2. Hypothesis:

Patients who show a bronchospasmolytic effect in their functional pulmonary test (FEV1 increased by at least 5%) within four hours of taking montelukast also show a positive response (defined as a combination of at least two variables (see section on the definition of responders/non-responders during treatment)) after 12 weeks of treatment. Conversely, patients who show no acute effect do not have a positive response during long-term therapy.

In other words, the results of the acute pharmacologic effect correspond to the effect during long-term therapy.

5. Aim of the study:

The main aim of the study is to develop a method that allows responders to be distinguished from non-responders before long-term treatment is initiated. Subsidiary aims are to record changes in pulmonary functional parameters, NO concentrations and peak flow variability, the use of beta2 sympathomimetics and the asthma symptom score.

6. Patient selection:

The study will include approximately 30 patients aged 6 to 14 years with diagnosed bronchial asthma who have been on constant anti-inflammatory therapy for at least four weeks (GINA classes 2 and 3).

7. Study design:

This investigation is a single-center, two-phase, single-arm study. In order to detect a potential placebo effect, the treatment phase will be preceded by a single-blinded two-week placebo run-in phase, followed by a 12 week open-label treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with symptomatic bronchial asthma despite ongoing therapy
* Age 6-14 years
* Asthma diagnosed at lease six months previously (by a special pulmonary allergologic outpatient unit)
* Demonstration of reversibility (FEV1 increased by at least 12% after bronchospasmolysis with a beta2 sympathomimetic). This can be determined at the screening visit or within the previous three months.
* Patients who are either steroid-naive or who received constant doses of the following medi¬cations within the previous four weeks:

  * Beclomethasone dipropionate: up to 400 µg daily
  * Fluticasone propionate: up to 200 µg daily
  * Budesonide: up to 400 µg daily
* Patients who are able to reliably complete the asthma diary and perform peak flow measurements according to instructions.
* Girls of childbearing potential must have acceptable methods of contraceptions, including sexual abstinence.

Exclusion Criteria:

* Patients who were treated with systemic steroids within the previous 30 days
* Patients using one of the following asthma medications:

  * Systemic steroids
  * Nedocromil, DNCG
  * Theophylline
  * Ketotifen
  * Systemic or long-acting beta2 sympathomimetics
* Patients who have experienced one of the following events within the previous 30 days:

  * A change in asthma medication
  * Pulmonary infection
  * Hospitalization due to bronchial asthma or any other respiratory condition
* Patients who are currently participating in another clinical trial or have done so within the previous 30 days.
* Patients known or expected to react hypersensitively to components of the investigational medication
* Patients receiving Phenobarbital, Phenytoin, Rifampicin (medications that are metabolized by Cytochrom P450
* Patients with analgetic intolerance
* Pregnant females

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Patients who show a bronchospasmolytic effect in their functional pulmonary test (FEV1 increased by at least 5%) within four hours of taking montelukast. | 14 days after run in

SECONDARY OUTCOMES:
symptom score, PEAK-Flow, rescue medication, exhaled NO | 2 weeks after run in and 14 weeks after run in

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA VON BERG, MD, Principal Investigator — Marien Hospital Wesel; FORSCHUNGSINSTITUT ZUR PRÄVENTION VON ALLERGIEN UND ATEMWEGSERKRANKUNGEN IM KINDESALTER AN DER kLINIK FÜR KINDER UND JUGENDMEDIZIN
Locations (1):
- Marien Hospital Wesel gGmbH, Wesel, North Rhine-Westphalia, Germany